CLINICAL TRIAL: NCT03933527
Title: The Effect of Staining Beverage on Color Alteration During In-office Tooth Bleaching: A Randomized Controlled Clinical Trial.
Brief Title: The Effect of Staining Beverage on Color Alteration During In-office Tooth Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Hao Yu, Fujian Medical University, Fujian Medical University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 20190214
Record Dates: First submitted 2019-04-27; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Tooth Discoloration
Keywords: tooth bleaching; staining beverage
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: factorial assignment
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Participants will receive in-office tooth bleaching with 40% hydrogen peroxide (Opalescence Boost PF 40%) for the maxillary anterior teeth (2 sessions, with a 1-week interval).
- coffee group (Experimental): Participants will receive in-office tooth bleaching with 40% hydrogen peroxide (Opalescence Boost PF 40%) for the maxillary anterior teeth (2 sessions, with a 1-week interval).During the tooth bleaching procedure and 3 weeks after the procedure,the participants will be instructed to make coffee rinses for 30 seconds, four times daily.
  Interventions: Behavioral: making staining beverage rinse during in-office tooth bleaching
- tea group (Experimental): Participants will receive in-office tooth bleaching with 40% hydrogen peroxide (Opalescence Boost PF 40%) for the maxillary anterior teeth (2 sessions, with a 1-week interval).During the tooth bleaching procedure and 3 weeks after the procedure,the participants will be instructed to make tea rinses for 30 seconds, four times daily.
  Interventions: Behavioral: making staining beverage rinse during in-office tooth bleaching

INTERVENTIONS:
Behavioral: making staining beverage rinse during in-office tooth bleaching — the subjects in experimental group should make staining beverage(coffee or tea) rinse for 30 second, four times daily.
  Arms: coffee group; tea group

SUMMARY:
This double-blind randomized controlled clinical trial aimed to investigate the effect of staining beverage on color alteration of in-office tooth bleaching procedures.

DETAILED DESCRIPTION:
Sixty-three eligible participants (25 males and 38 females, mean age 26.5 years) with at least one maxillary tooth demonstrating shade A3 or darker will be recruited and randomly allocated into 3 groups (n = 21), according to the different staining beverage used in this clinical trial: Coffee for group C, Tea for group T, and distilled water for group W. All participants will receive in-office tooth bleaching with 40% hydrogen peroxide (Opalescence Boost PF 40%) for the maxillary anterior teeth (2 sessions, with a 1-week interval). The participants will be instructed to use only the provided beverage rinses for 30 seconds, four times daily. Colour parameters (CIE L*, a*, b*) will be measured with a spectrophotometer (Vita Easyshade Advance 4.0) at baseline (T1), after the first bleaching session (T2), after the second bleaching session (T3), 1 week after the completion of in-office bleaching (T4), and 3 weeks after the completion of in-office bleaching (T5). The colour differences (ΔE) and whiteness index (W) will also be calculated. The data will be statistically analysed through repeated ANOVA and Tukey's test (α = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* patients between 18 and 30 years of age, with fully erupted upper and lower incisors and canines without dental or periodontal disease or restorations, and with at least one maxillary tooth presenting color score A3 or darker, as measured with the Vita Classical guide (Vita Zahnfabrik, Bad Sa ̈ ckingen, Germany) ordered by brightness

Exclusion Criteria:

* patients with systemic diseases or oral mucosal disorders, previous bleaching treatment, patients undergoing orthodontic treatment, pregnant women, people with known allergy to the product ingredients, smokers, and alcohol abusers.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Change in tooth colour | 4 weeks
  Colour parameters (CIE L*, a*, b*) will be measured with a spectrophotometer (Vita Easyshade Advance 4.0). The color alteration after each session will be given by the differences between the values obtained at the sessions and the baseline (∆E).

SECONDARY OUTCOMES:
Change in tooth whiteness | 4 weeks
  The whiteness index will be registered at the sessions and the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yu, Principal Investigator — Fujian Medical University, China
Locations (1):
- Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen YH, Yang S, Hong DW, Attin T, Yu H. Short-term effects of stain-causing beverages on tooth bleaching: A randomized controlled clinical trial. J Dent. 2020 Apr;95:103318. doi: 10.1016/j.jdent.2020.103318. Epub 2020 Mar 10. PMID 32169479